## Official Title: EngagINg the COmmunity to Reduce Preterm Birth Via Adherence To an Individualized Prematurity Prevention Plan (INCORPorATe IP3)

NCT: NCT04933812

IRB Document Date: 01/17/2023

Previous studies have shown preterm births (PTB) are high in non-Hispanic Black (NHB) women and women are more likely to have a PTB if they previously had one. Pregnant women with history of PTB at Duke Maternal Fetal Medicine receive IP3 plans to reduce the risk of recurrent PTB and these interventions are often stressful. The EnagagINg the Community to Reduce Preterm Birth via Adherence To an Individualized Prematurity Prevention Plan (INCORPorATe IP3) was developed to provide support for NHB women who had prior PTB. This intervention included information provided through Facebook group discussions with doulas and Zoom group meetings to review a variety of pregnancy-related topics.

Participants received questionnaires to complete at intake, between 20-28 weeks GA, and after 30 weeks GA in addition to group satisfaction surveys after each Zoom meeting. Results from the questionnaires and surveys will be reported as counts (percentages) for categorical variables and mean (SD), median (IQR), and range for continuous variables.

| Table 1. Participant Characteristics | |
|---|---|
| Characteristic | |
| Age (mean, SD) | |
| Number of Prior Preterm Births (median, IQR) | |
| Insurance Status | |
| Public | |
| Private | |
| None | |
| Body mass index at prenatal care intake (mean, SD) | |
| Chronic hypertension | |
| Pre-gestational Diabetes | |
| Tobacco use at any time in pregnancy | |
| Preterm Birth Preventative Recommend | ations (i.e., IP3 plan) |
| Lifestyle modifications (n, %) | |
| Cervix length/Cerclage (n, %) | |
| Progesterone (n, %) | |
| Low Dose Aspirin (n, %) | |
| All data are reported as n (%) unless detailed otherwi | ise |

| Table 2. Feasibility and Acceptability Measures |
|-------------------------------------------------------------|
| Recruitment: |
| #Eligible people approach/ # recruited |
| Facebook Engagement: |
| Number of participants who logged onto the Facebook page |
| Number of participants who posted/reposted anything |
| Facebook engagement metrics |
| Group Social Support (GSS) Session Engagement: |
| Median number of GSS visits attended [IQR] |
| Number (%) of participants who attending 5 or more sessions |

| Table 3. Gro | Table 3. Group Social Support Sessions | | | |
|---|---|---|---|---|
| Session # | Topics Covered | # Attended/#<br>Enrolled at<br>session<br>timepoint | Post-meeting survey<br>% very satisfied<br>% somewhat satisfied<br>%non satisfied | No-Show Survey Results |
| #1 | | | | |
| Date | | | | |
| #2<br>Date | | | | |
| #3 | | | | |
| Date | | | | |
| #4 | | | | |
| Date | | · | | |
| #5 | | | | |
| Date | | | | |
| #6 | | | | |
| Date | | | | |
| 40.000 | | | | |
| **** | | | | |

| #0 | | . ' | | | |
|---|---|---|---|---|---|
| Date | | | | | |
| | | | | | 7 |
| | *************************************** | | | | e-manual . |
| | - House the same that the same | Photos III and the second state of the second | | <br> | _ |
| | Feasibility and Accep | stability Measures | | | |
| Recruitment: | | | | | |
| #eligible people | approach/#recruit | .ed | | | |
| Retention: | | | | | |
| # participants w | ho completed all su | rvey measures | | | |
| Avg # survey me | easures completed/p | participant | | | |
| Facebook Engag | gement: | A. Control of the Con | | | |
| Number of parti | icipants who logged | onto the Facebook | page | | |
| Number of parti | icipants who posted, | /reposted anything | | | |
| Facebook engag | | , - | | | |
| Healthcare Utiliz | | | | | 7 |
| 7,00,0,00,00 | | | | <br> | 7 |
| | - | | | | _ |

| Table 5. Adherence and Pregnancy Outcomes | |
|---|---|
| Preterm Birth Preventative Recommendation Adherence (adhe | ered/recommended, percent) |
| Lifestyle Modifications | |
| IOM weight gain guidelines | |
| Tobacco cessation | |
| Supplemental Progesterone | |
| 17-P | |
| Vaginal progesterone | |
| Cerclage/Serial Cervix Length | |
| Cerclage | |
| Serial cervix lengths | |
| Low Dose Aspirin | |
| Pregnancy Outcomes (n, %) | |
| Preterm Birth/Gestational Age Outcomes: | |
| Preterm delivery <37 weeks | |
| Gestational age at delivery in weeks, mean (SD) | |
| Length of gestation in current pregnancy compared to earliest | |
| preterm birth, mean (SD) | |
| Maternal Outcomes: | |
| Preeclampsia/gestational hypertension | |
| Number of antepartum triage evaluations, median (IQR) | |
| Antepartum hospital admission | |
| Length of delivery admission in days, median (IQR) | |
| Neonatal Outcomes: | |
| Birth weight in grams, mean (SD) | |
| Neonatal Intensive care unit admission | |

| Table 6. Secondary Quantitative Measure (mean, SD) | Intake<br>N= 32 | Protocol<br>Completion<br>N= | Change |
|---|---|---|---|
| Interpersonal Process of Care (IPC-18) at protocol completion<br>Description: Validated 18-question instrument that measures patient care expeach domain range from 1 to 5 on a Likert scale | perience during clin | ical visits in four domains | . Scores for |
| Communication Domain | | | |
| Lack of clarity (higher scores are negative, donate increased lack of clarity from clinicians) | | | |
| Elicits concern (higher scores are positive, denotes the clinician elicited concerns more often) | | | |
| Explain results (higher scores are positive, denotes the clinician explained results more often) | | | |
| Decision Making Domain | | | |
| Decision Making (higher scores are positive, denoting more collaborative decision making between the clinician and patient) | | | 7. 110. 1110. |
| Interpersonal Style Domain | | | |
| Emotional support (higher scores are positive, denoting more emotional support from the clinician) | | | |
| Discrimination due to race/ethnicity (higher scores are negative, donate increased discrimination from clinicians) | | | 400 |
| Disrespectful to office staff (higher scores are negative, donate increased disrespectful behavior from clinicians towards office staff) | | | |
| Maternal Social Support Scale (MSSS) Description: Six question questionnaire answered from 1 to 5 on a Likert scale MSS at intake | , higher scores are | positive and denote incre | ased support |
| MSSS at protocol completion | | | |
| Pregnancy Specific Anxiety (PSA) at 28 weeks | | | |
| Description: Frequency of four emotions rated from 1 to 5 on a Likert scale, hi | gher scores are neg | ative and denote incress | ed anviety |
| PSA at intake | Bile i beores die Heg | daye and denote increas | cu anxiety |
| PSA at 3 <sup>rd</sup> trimester | | | |